CLINICAL TRIAL: NCT01602731
Title: Targeted Intervention to Improve Medication Adherence in Cognitively Impaired Patients With Heart Failure
Brief Title: Targeted Intervention to Improve Medication Adherence in Cognitively Impaired Patients With HF (TARGET)
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RRP 12-198
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: medication adherence
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Automated Medication Dispensing Device (Experimental): Subjects with <88% medication adherence, determined by 30-day pillcount, and with cognitive impairment (determined by Saint Louis University Mental Status score) proceeded to AMDD portion of study.
  Interventions: Device: Automated Medication Dispensing Device

INTERVENTIONS:
Device: Automated Medication Dispensing Device — All patients had a pre-filled medication dispensing machine set up at their homes, filled by home health nurses once a month. Safety phone call was made by the AMDD company if doses were missed.
  Other Names: AMDD

SUMMARY:
Trialing an automated medication dispensing device (AMDD) to improve medication adherence in patients with heart failure.

DETAILED DESCRIPTION:
Background:

Medication adherence [MA] is a complex issue depending on both patient and healthcare factors. Non-adherence due to patient-dependent factors is common; analyses of large broad-based clinical trials in the general population demonstrate that 20-30% of study medication doses may be missed. In community-dwelling HF patients with polypharmacy this percentage is likely even higher. One of the factors in poor adherence in elderly non-HF patients has been shown to be cognitive impairment [CI]. Non-adherence to medical regimen is one factor that is associated with worse outcomes in patients with HF, including readmissions. Measures that improve MA are also likely to improve outcomes.

Objectives:

We evaluated a novel intervention incorporating new technology with the goal of improving adherence in patients with HF and CI. Specific objectives of the study were (1) to assess the feasibility of using the Automated Medication Dispensing Device (AMDD) in veterans with HF and CI by measuring patient qualifying rate, consent rate, user rate, patient-level response rate, medication-level response rate, and success rate, (2) to calculate the improvement of MA based on pill counts before and after the introduction of the AMDD, and (3) qualitatively describe patient satisfaction with the AMDD and the reasons for not using the AMDD.

Methods:

This pilot was designed as a feasibility study testing an intervention using a commercially available, off the shelf Automated Medication Dispensing Device (AMDD) with subjects serving as their own controls. The study was conducted at the VALLHS, Loma Linda, CA which serves a population of 246,000 veterans. The study planned to enroll 50 patients with HF and CI (defined as SLUMS score of <27 in a person with high school education or <25 in a person with less than high school education) from the outpatient HF clinic. Baseline adherence to prescribed medications was measured by an initial 30-day pill count (month 1). Subjects with baseline adherence <88% were given the AMDD to use for 90 days (one month to familiarize the study subjects with the device, two months to collect outcome data). This dispenser was pre-filled by home health nurses once a month; the dispenser is equipped with an alarm mechanism that alerts the patient to take the medications; when the patient pushes the button on the device, it will dispense the medications. 30-day pill counts were performed while patients were using the AMDD on months 3 and 4. The study was powered to detect the success rate of the AMDD, defined as both patient acceptance and a clinical response to the AMDD.

Status:

Complete. This project was opened for recruitment as of July 1, 2012. The study is now closed for recruitment and all enrolled patients have completed the intervention. Manuscript outlining the findings of this study and discussing the available interventions to improve medication adherence is in progress.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of clinical heart failure
* English-speaking
* Able to provide informed consent
* Able to participate in cognitive function testing
* Age over 18

Exclusion Criteria:

* Life expectancy < 6 months
* Documented dementia requiring a caregiver
* inability to set up the AMDD at the patient's home due to technical limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helme Silvet, MD, Principal Investigator — VA Medical Center, Loma Linda
Locations (1):
- VA Medical Center, Loma Linda, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This project was opened for recruitment as of July 1, 2012. Enrollment for the study originally took place in the heart failure (HF) clinic and Investigator's circle of confidentiality, but after poorer than anticipated enrollment, screening was expanded to all outpatients at the VALLHS with a diagnosis of HF.
Groups:
- Automated Medication Dispensing Device: Subjects with <88% medication adherence, determined by 30-day pillcount, will proceed to AMDD portion of study
  Automated Medication Dispensing Device: A pre-filled medication dispensing machine with a safety phone call if doses are missed
Period: Overall Study
Arm/Group | Automated Medication Dispensing Device
Started | 45
Cognitive Impairment | 44 (After repeat cognitive testing, additional 1 patient had no cognitive impairment and did not proceed)
Poor Medication Adherence | 24 (24 out of 35 patients who completed 1-month pill counts had medication adherence <88%.)
Completed | 15
Not Completed | 30

BASELINE CHARACTERISTICS:
Groups:
- AMDD: Subjects with <88% medication adherence, determined by 30-day pillcount, will proceed to AMDD portion of study
  Automated Medication Dispensing Device: A pre-filled medication dispensing machine with a safety phone call if doses are missed
Arm/Group | AMDD
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 10
  White | 25
  More than one race | 9
  Unknown or Not Reported | 0
Education level [Number; unit: participants]
  no high school | 2
  high school or equivalent | 10
  some college | 23
  college degree | 7
  postgraduate degree | 3
Living arrangements [Number; unit: participants]
  live alone | 11
  live with others | 34
Saint Louis University Mental Status score [Mean (Standard Deviation); unit: units on a scale] — Saint Louis University Mental Status Score is measured on the scale of 30 and contains 11 questions that incorporate cognitive tasks. It has been validated in different studies and has high sensitivity and specificity in detecting dementia, as well as mild cognitive impairment. Score of <27 is in a person with high school education or <25 in a person with less than high school education is considered abnormal and consistent with cognitive impairment. The total range for the SLUMS scale could range from 1 (severe dementia) to 30 (normal).
  units on a scale | 20.9 (5.8)
Medication adherence [Mean (Standard Deviation); unit: Percentage] — Medication adherence was measured by 30-day pill counts and included all prescribed medications, except the ones prescribed on an as-needed basis. To capture both overtaking and undertaking medication, a "delta" was determined for each medication by computing the absolute difference between the number of pills taken and the number prescribed over the 30-day period. The delta values for each medication were summed for each individual subject, divided by the total number of pills prescribed, subtracted from 1, and finally multiplied by 100 to obtain an adherence score expressed as a percentage.
  Percentage | 69.9 (12)
Full Range of Saint Louis University Mental Status Scores [Mean (Full Range); unit: units on a scale] | 20.9 [14 to 28]

OUTCOME MEASURES:

1. Secondary Outcome: Efficacy of AMDD to Improve Medication Adherence
Description: Change in medication adherence (proportion of pills taken of prescribed, as measured by pillcount) after the implementation of the AMDD
Time Frame: 30-day pill count before the use of AMDD and with AMDD
Measure: Mean (Full Range); unit: percentage of adherence
Groups:
- Before AMDD: Adherence was measured by 30-day pill count before the use of AMDD
- After AMDD: Adherence was measured with the use of the AMDD as a 30-day pill count
Arm/Group | Before AMDD | After AMDD
Number analyzed (Participants) | 15 | 15
percentage of adherence | 65 [30 to 83] | 97 [91 to 100]

2. Primary Outcome: Feasibility of AMDD to Improve Medication Adherence Via Completion Rate
Description: Rate that patient population completed set-up of AMDD was evaluated quantitatively.
Time Frame: 4 months
Population: Of 45 patients who started the study, 24 patients met the predetermined criteria for AMDD. Though all of the patients had agreed to set up the AMDD in their home, only 15 out of 24 ended up completing the setup in their home.
Measure: Number; unit: participants
Arm/Group | Automated Medication Dispensing Device
Number analyzed (Participants) | 45
participants | 15

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the intervention part of the study (4 month-period for each patient).
Description: We did not collect data on patient outcomes or hospitalizations because the study did not use investigational medications or devices, and only tested feasibility of a patient self-care assist device. We did collect data on the technical support for the medication dispensing device, as well as technical issues with the device.
Arm/Group | AMDD
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
Low enrollment in the study reflects the fact that many patients with HF do not admit the need for assistance with their medications. Patients should first be tested for the presence of cognitive impairment and baseline medication adherence problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No